CLINICAL TRIAL: NCT07366099
Title: Application of Al18F-NOTA-LM3 PET/CT in the Diagnosis and Evaluation of Tumor-Induced Osteomalacia
Brief Title: Al18F-NOTA-LM3 PET/CT in Patients With TIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALFLM3TIO
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: Tumor-Induced Osteomalacia
MeSH Terms: conditions — Oncogenic osteomalacia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-LM3 and 68Ga-DOTATATE PET/CT scan (Experimental): Patients of TIO PET/CT imaging: Patients will perform an Al18F-NOTA-LM3 PET/CT as well as a 68Ga-DOTATATE PET/CT.
  Interventions: Drug: Diagnostic Test: Al18F-NOTA-LM3; Drug: Diagnostic Test: 68Ga-DOTATATE

INTERVENTIONS:
Drug: Diagnostic Test: Al18F-NOTA-LM3 — Al18F-NOTA-LM3 will be injected into the patients. Patients will undergo a whole-body PET/CT scan 60-120 minutes after injection.
Drug: Diagnostic Test: 68Ga-DOTATATE — 68Ga-DOTATATE will be injected into the patients. Patients will undergo a whole-body PET/CT scan 40-60 minutes after injection.

SUMMARY:
This is a pilot study to assess the value of whole-body Al18F-NOTA-LM3 PET/CT in patients with tumor-induced osteomalacia.

DETAILED DESCRIPTION:
Tumor-induced osteomalacia (TIO) is a rare paraneoplastic syndrome. The main cure for TIO is surgical removal of the responsible tumor. Somatostatin receptors (SSTR) targeted PET imaging with radiolabeled somatostatin analogs can help locate these tumors. It can detect culprit tumors in TIO patients, even small ones that CT or MRI might miss. 68Ga-DOTATATE is the most commonly used SSTR PET tracer for TIO, recommended as the first-line imaging tool to find the causative tumor.

Compared to 68Ga-based tracers, 18F-labelled radiotracers offer several advantages, including higher cyclotron production, lower positron energy, and longer half-life. These features may improve image quality. Al18F-NOTA-LM3 is an SSTR2 specific antagonist used as a PET tracer. This pilot study is designed to compare Al18F-NOTA-LM3 with 68Ga-DOTATATE in the same group of TIO patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* Suspected or confirmed TIO patients.

Exclusion Criteria:

* Combined with other types of tumors.
* Severe liver or renal dysfunction (ALT/AST≥5 ULN, GFR<30ml/min).
* Pregnant or breast-feeding women.
* Inability to perform PET/CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | From study completion to 6 months after completion.
  Sensitivity and specificity of Al18F-NOTA-LM3 PET/CT for TIO in comparison with 68Ga-DOTATATE PET/CT

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | From study completion to 6 months after completion.
  Compare the SUVmax of tumor derived from Al18F-NOTA-LM3 and 68Ga-DOTATATE PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China